CLINICAL TRIAL: NCT04926207
Title: SIT Less! Interrupting Prolonged Sitting With Brief Physical Activity Bouts to Improve Neurocognitive Function in Adults With Obesity
Brief Title: The Effects of Interrupting Prolonged Sitting With Bouts of Physical Activity on Neurocognitive Function in Obesity
Acronym: SITLess
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20633
Record Dates: First submitted 2021-05-24; First posted 2021-06-15 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Obesity
Keywords: Sedentary Behavior; Executive Function; Event Related Potentials; Insulin; Glucose
MeSH Terms: conditions — Obesity; Sedentary Behavior; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Breaks Intervention (Experimental): Participants will sit continuously for 3 hours and interrupt their sitting by walking on a treadmill at a moderate intensity for 3 min.
  Interventions: Behavioral: Physical Activity Breaks Intervention
- Talking Breaks Control (Active Comparator): Participants will sit continuously for 3 hours. They will interrupt solitary sitting activities (while remaining seated) by talking to a researcher for 3 min on pre-selected topics of general interest.
  Interventions: Behavioral: Talking Breaks Control

INTERVENTIONS:
Behavioral: Physical Activity Breaks Intervention — Participants will be asked to walk on a treadmill for 3 min at a moderate intensity (55% of heart rate reserve) at an increasing speed and incline to reach and maintain their target heart rate.
  Arms: Physical Activity Breaks Intervention
Behavioral: Talking Breaks Control — Every 30 min a researcher will start a brief conversation with a participant based on a pre-selected topic, which will change with each break. Topics are standardized across participants and include, for example, pollution, smart clothes, and hydration. A presentation will be followed by questions and answers. The break will last 3 min.
  Arms: Talking Breaks Control

SUMMARY:
It is projected that by 2030 almost 50% of adults in the USA will have obesity. High sedentariness and physical inactivity contribute to the obesity pandemic. Neurocognitive deficits compound the global burden of obesity. Specifically, adults with obesity underperform on tasks of executive functioning, which underpin goal-directed behavior and have been linked to occupational success. Growing evidence suggests poorer executive functioning among more sedentary adults. Emergent studies have shown that accumulating sedentary time in prolonged bouts (e.g., remaining sedentary continuously 20 min or more) may decrease the ability to control distractions along with working memory. Interrupting prolonged sitting with brief bouts of physical activity is an effective strategy to improve postprandial glucose metabolism. However, the effects of this simple intervention on neural processes supporting executive functioning remain unknown. Accordingly, the aim of this study is to test the effects of interrupting prolonged sitting with frequent (every 30 min) but brief (3 min) physical activity bouts on inhibitory control, working memory, and their neuroelectric indices (N2, P3a, and P3b components of event-related brain potentials). Our secondary aim is to explore the potential mechanisms underlying the effects of interrupting prolonged sitting with physical activity on cognitive and brain function through glucose metabolism and insulin physiology. Findings from this study will help advance our understanding of how restructuring sedentary time may help improve cognitive and brain functions among adults with obesity.

DETAILED DESCRIPTION:
Measurements of cognitive and brain function will be taken before, and after three hours of prolonged sitting. Metabolic, heart rate, and blood pressure measures, along with the ratings of fatigue will be collected before and during the three-hour prolonged sitting time. The prolonged sitting time will be either interrupted with physical activity breaks or with sedentary breaks (attention control). Habitual physical activity, sedentary behavior, sleep, and dietary intake will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* • Informed consent

  * Age 21-64 years
  * BMI within ≥ 30 and < 40 kg/m2 range
  * Pre-menopausal
  * Fasting plasma glucose (FPG) < 100 mg/dL
  * Resting blood pressure: systolic < 160 mmHg or diastolic < 100 mmHg
  * Employed in sedentary occupation (i.e., participants reporting sitting on average 6 h/d on a weekday and with objectively assessed sitting time ≥ 8 h/day)
  * Physically inactive (i.e., engaging in < 150 min of moderate or < 75 min of vigorous or any combination of the two intensities per week)
  * Participants must have had no prior diagnosis of cognitive or physical disability (e.g., ADHD, severe asthma, epilepsy, chronic kidney disease, or dependence upon a wheelchair/walking aid)
  * Free of medication that could affect cognitive function or metabolism
  * Normal or corrected-to-normal vision based on the minimal 20/20 standard in order to complete the cognitive task (below 20/20 vision)
  * Must be able to engage in vigorous exercise
  * Fluency in English

Exclusion Criteria:

* • Impaired glucose tolerance defined as fasting plasma glucose (FPG) < 100 mg/dL

  * Oral glucose tolerance test (OGTT) blood glucose values ≥ 200 mg/dL
  * Participants with any psychiatric, neurological or metabolic disorder
  * Participants who have or are currently taking the medication that could affect cognitive function, metabolism or weight status
  * Participants with substance abuse
  * Participants with a standardized score on the test of general cognitive abilities below 85
  * Participants with anemia
  * Pregnant women or those with a possible pregnancy
  * History of injury to the spinal cord

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Neuroelectric measures of inhibitory control - P3 component of event-related potentials (ERPs) | Assessed immediately before and after the intervention (on the same day as intervention)
  The change in the P3 component measured during the modified flanker task
Neuroelectric measures of inhibitory control - N2 component of event-related potentials (ERPs) | Assessed immediately before and after the intervention (on the same day as intervention)
  The change in the N2-ERP component measured during the modified flanker task.
Inhibitory control measured with a modified flanker task - accuracy | Assessed immediately before and after the intervention (on the same day as intervention)
  The change in accuracy on the modified flanker task
Inhibitory control measured with a modified flanker task - reaction time | Assessed immediately before and after the intervention (on the same day as intervention)
  The change in measures of reaction time on the modified flanker task
Neuroelectric measures of working memory - P3-ERP component | Assessed immediately before and after the intervention (on the same day as intervention)
  The change in the P3-ERP component during the n-back task.
Working memory measured with an n-back task - accuracy | Assessed immediately before and after the intervention (on the same day as intervention)
  The change in accuracy on the n-back task
Working memory measured with an n-back task - reaction time | Assessed immediately before and after the intervention (on the same day as intervention)
  The change in measures of reaction time on the n-back task

SECONDARY OUTCOMES:
Post-prandial insulin response during an oral glucose tolerance test | Assessed during the intervention
  Insulin Area Under the Curve (AUC)
Post-prandial glucose response during an oral glucose tolerance test | Assessed during the intervention
  Glucose Area Under the Curve (AUC)
Matsuda index | Assessed during the intervention
  Insulin Sensitivity measured with Matsuda index
Stumvoll metabolic clearance rate (MCR) | Assessed during the intervention
  Insulin Sensitivity expressed as Stumvoll metabolic clearance rate

CONTACTS AND LOCATIONS:
Overall Officials: Dominika M Pindus, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No